CLINICAL TRIAL: NCT06579287
Title: A Phase II Study to Determine the Safety and Efficacy of SHJ002 Sterile Ophthalmic Solution on Myopia Control in Subjects Aged 3-12 Years.
Brief Title: A Study of SHJ002 Sterile Ophthalmic Solution for Myopia Control
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunhawk Vision Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHJ002-MY201
Record Dates: First submitted 2024-08-15; First posted 2024-08-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Myopia, Progressive
Keywords: Myopia
MeSH Terms: conditions — Myopia, Degenerative; Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SHJ002 (Experimental): The assigned eyedrops will be instilled in both eyes once per day, one drop per application, 7 days a week, for 52 weeks.
  Interventions: Drug: SHJ002
- Atropine (Active Comparator): The assigned eyedrops will be instilled in both eyes once per day, one drop per application, 7 days a week, for 52 weeks.
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: SHJ002 — Topical ophthalmic
  Arms: SHJ002
Drug: Atropine — Topical ophthalmic
  Arms: Atropine

SUMMARY:
The objective of this study is to explore the safety and efficacy of SHJ002 Sterile Ophthalmic Solution relative to atropine in myopia control

SHJ002 is an antisense oligonucleotide to neutralize a specific microRNA.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female, age 3-12 years (inclusive).
2. Cycloplegic sphere of -1.00 D or worse in both eyes
3. Able to complete all study assessments and comply with the protocol
4. Literate or able to orally communicate.
5. Parent or guardian able and willing to provide written informed consent
6. Parent or guardian able and willing to assure subject compliance with the protocol, follow study instructions, and attend study visits
7. Able to tolerate eye drops in both eyes.
8. Be able and willing to avoid all disallowed medications and refractive correction
9. For female subjects of childbearing potential (those who have experienced menarche and who are not surgically sterilized [bilateral tubal ligation, hysterectomy, or bilateral oophorectomy]), a negative urinary test.
10. Women of childbearing potential must agree to use two reliable methods of contraception
11. Males not naturally or surgically sterile, who have a female partner of childbearing potential, must agree to use two reliable methods of contraception

Exclusion Criteria:

1. Axial length > 26 mm
2. Anisometropia
3. Astigmatism > 2.00 D
4. Intraocular pressure > 21 mm Hg or < 6 mm Hg
5. Active or recent history of severe ocular infection or inflammation
6. Previous incisional or laser surgery
7. Any clinically significant finding on slit lamp biomicroscopy or ophthalmoscopy

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of the cycloplegic spherical equivalent (SE) | from baseline visit to the final visit, up to 52 weeks

SECONDARY OUTCOMES:
Change of axial length | from baseline visit to the final visit, up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (9):
- Pacific Center for Advanced Vision Care Tanasbourne Vision Center, Hillsboro, Ohio, United States
- Taiwan (8):
  - Changhua Christian Hospital, Chang-hua
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Cung Memorial Hospital-Tucheng, New Taipei City
  - MacKay Memorial Hospital-Tamsui, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No